CLINICAL TRIAL: NCT01432665
Title: Lybrido for Female Sexual Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emotional Brain NY Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EB82
Record Dates: First submitted 2011-08-17; First posted 2011-09-13 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Sildenafil Citrate; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Experimental): 30 subjects administered a placebo
  Interventions: Drug: Placebo
- sildenafil + testosterone combination drug 1 (Experimental): 30 subjects are given combination drug 1 (sildenafil 25mg and testosterone 0.25mg)
  Interventions: Drug: Sildenafil; Drug: Testosterone
- Sildenafil and testosterone combination drug 2 (Experimental): Sildenafil 50mg and testosterone 0.25mg
  Interventions: Drug: Sildenafil; Drug: Testosterone
- Sildenafil and testosterone combination drug 3 (Experimental): 30 subjects are given sildenafil 25mg and testosterone 0.50mg
  Interventions: Drug: Sildenafil; Drug: Testosterone
- Sildenafil and Testosterone Combination drug 4 (Experimental): 30 subjects are given sildenafil 50mg and testosterone 0.50mg
  Interventions: Drug: Sildenafil; Drug: Testosterone
- Sildenafil 50mg (Experimental): 30 subjects are given sildenafil 50mg
  Interventions: Drug: Sildenafil
- Testosterone 0.50mg (Experimental): 30 subjects are given testosterone 0.5mg
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Placebo — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Placebo
Drug: Sildenafil — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Sildenafil 50mg; Sildenafil and Testosterone Combination drug 4; Sildenafil and testosterone combination drug 2; Sildenafil and testosterone combination drug 3; sildenafil + testosterone combination drug 1
Drug: Testosterone — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Sildenafil and Testosterone Combination drug 4; Sildenafil and testosterone combination drug 2; Sildenafil and testosterone combination drug 3; Testosterone 0.50mg; sildenafil + testosterone combination drug 1

SUMMARY:
The Lybrido study is a double-blind, randomized, placebo-controlled study with a 4-week baseline establishment period, 16 week treatment period and a follow up period for a total of 26 weeks on study. Subjects are randomly to one of seven treatment arms. The study investigates the effective dose of Lybrido in increasing the number of satisfactory sexual episodes in the domestic setting in 210 healthy female subjects with hypoactive sexual desire disorder and low sensitivity for sexual cues (30 subjects per group).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Female 21 to 70 years of age, inclusive, pre- or postmenopausal, with HSDD (comorbidity with female sexual arousal disorder and/or female orgasmic disorder [FOD; only as secondary diagnosis] is allowed). The diagnosis of HSDD will be established by a trained professional.
3. Low sensitivity for sexual cues
4. Be involved in a stable relationship and have a partner who will be at home for the majority of the study duration
5. Healthy according to normal results of medical history, physical examination, laboratory values, and vital signs; exceptions may be made if the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

1. Any underlying cardiovascular condition, including unstable angina pectoris, that would preclude sexual activity
2. History of myocardial infarction, stroke, transient ischemic attack, or life-threatening arrhythmia within the prior 6 months
3. Uncontrolled atrial fibrillation/flutter at screening or other significant abnormality observed on electrocardiogram (ECG)
4. Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure > 90 mmHg. For subjects > 60 years old and without diabetes mellitus, familial hypercholesterolemia, or cardiovascular disease: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure > 90 mmHg
5. Systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg
6. Use of oral contraceptive containing anti-androgens
7. Use of oral contraceptive containing 50 μg estrogen or more
8. Positive test result for Chlamydia or gonorrhea
9. Pregnancy or intention to become pregnant during this study (Note: A urine pregnancy test will be performed in all women prior to the administration of study medications.)
10. Lactating or delivery in the previous 6 months
11. Significant abnormal pap smear in the previous 12 months
12. History of bilateral oophorectomy
13. Other unexplained gynecological complaints, such as clinically relevant abnormal uterine bleeding patterns
14. Liver and/or renal insufficiency (aspartate aminotransferase and alanine aminotransferase > 3 times the upper limit of normal and/or glomerular filtration rate < 29 mL/min based on the Cockcroft and Gault formula)
15. Current clinically relevant endocrine disease or uncontrolled diabetes mellitus
16. Current clinically relevant neurological disease which, in the opinion of the investigator, would compromise the validity of study results, or which could form a contraindication for sildenafil and/or testosterone use
17. History of hormone-dependent malignancy
18. Vision impairment, such as partial or complete blindness or color blindness
19. Dyslexia
20. Positive test result for human immunodeficiency virus, hepatitis B, or hepatitis C (acute and chronic hepatitis infection)
21. History of (childhood) sexual abuse that, in the opinion of the investigator, could have negative psychological effects when testosterone is administered
22. (Treatment for) a psychiatric disorder that, in the opinion of the investigator, would compromise the validity of study results or which could be a contraindication for sildenafil and/or testosterone use
23. Current psychotherapeutic treatment for female sexual dysfunction
24. Current sexual disorder of vaginismus or dyspareunia according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (text revision).
25. A substance abuse disorder that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study (Mild or moderate alcohol consumption is allowed but must be stopped 12 hours before the home measurement [Stroop task].)
26. Positive test result for illicit drugs
27. Use of potent CYP3A4 inhibitors (eg, ritonavir, ketoconazole, itraconazole clarithromycin, erythromycin and saquinavir)
28. Use of potent CYP3A4 inducers (eg, carbamazepine, phenytoin, phenobarbital, St John"s wort, rifampin)
29. Use of nitrates or nitric oxide donor compounds
30. Use of selective serotonin reuptake inhibitors, tricyclic antidepressants, or other antidepressants
31. Use of any other medication that interferes with study medication (eg, monoamine oxidase [MAO] inhibitors [includes classic MAO inhibitors and linezolid])
32. Use of medication (including herbs) that would compromise the validity of study results
33. Use of testosterone therapy within 6 months before study entry
34. Illiteracy, unwillingness, or inability to follow study procedures
35. Participation in other clinical trials within the last 30 days
36. Any other clinically significant abnormality or condition which, in the opinion of the investigator, might interfere with the participant"s ability to provide informed consent or comply with study instructions, compromise the validity of study results, or be a contraindication for sildenafil and/or testosterone use

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The number of satisfactory sexual encounters based on event questionnaires on active drug as compared to placebo during double-blind treatment period episodes in the domestic setting. | 20 weeks
  Efficacy is estimated by self reporting by subjects using daily event questionnaires, recorded within 24 hours after a sexual event. The number of events between a 4-week baseline establishment period will be compared with the number of events during the 8 week double-blind treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.

SECONDARY OUTCOMES:
Sexual satisfaction | 20 Weeks
  Sexual satisfaction will be evaluated based on a global satisfaction assessment comparing the 4-week establishment period with the 8 week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.
Sexual desire and arousal | 20 Weeks
  Sexual desire and arousal will be evaluated based on the 'desire' and 'arousal' domains of the Sexual Anamnesis Questionnaire, the Sexual Function questionnaire and weekly diaries throughout the course of the study.
Sexual motivation and inhibition | 20 Weeks
  Sexual motivation and inhibition will be assessed using the Sexual Motivation Questionnaire and comparing sexual motivation and inhibition between the 4-week establishment period and the 8-week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.
Safety and toleration | 20 Weeks
  Safety will be evaluated by: 1) AEs [Number of patients reporting AEs, number of patients reporting drug related AEs] 2)SAE [Number of patients reporting SAEs, number of patients reporting drug related SAEs]and 3) Changes in laboratory safety data [Number of patients reporting abnormal lab safety data, number of patients reporting drug related abnormal lab safety data]. These will be evaluated throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - San Diego Sexual Medicine, San Diego, California
  - The Center for Vulvovaginal Disorders, Washington D.C., District of Columbia
  - Meridien Research, Brooksville, Florida
  - Segal Institute Women's Health Clinic, North Miami, Florida
  - Compass Research, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Annapolis Sexual Wellness Center, Annapolis, Maryland
  - Maryland Prime Care Physicians, Stevensville, Maryland
  - Center for Sexual Medicine at Sheppard Pratt, Townson, Maryland
  - Women's Health Research Center, Plainsboro, New Jersey
  - Michael A. Werner, MD PC, Purchase, New York
  - Philadelphia Clinical Research, Philadelphia, Pennsylvania